CLINICAL TRIAL: NCT06899048
Title: Residual Paralysis in the Post Anesthesia Care Unit: The Association Between Residual Neuromuscular Block Risk Prediction Score and the Train-of-Four Ratio. A Prospective Single-Center Open-Label Cohort Study
Brief Title: The Association Between Residual Neuromuscular Block Risk Prediction Score and the Train-of-Four Ratio
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Faisal, Dr, Assiut University
Other Study IDs: 04-2025-201158
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-10

CONDITIONS: Muscle Relaxants
MeSH Terms: conditions — Muscle Hypotonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: residual neuromuscular block risk prediction score — it is a clinical tool designed to estimate the likelihood of residual neuromuxcular blockade in postoperative patients

SUMMARY:
evaluate the degree of association, and the predictive accuracy of the REPS (as a predictive tool) compared with the TOFr as a quantitative assessment tool for (rNMB) in surgical patients in the early postoperative phase. The TOFr will be measured at 0, 15, 30, 45, and 60 min after extubation.

ELIGIBILITY:
Inclusion Criteria:

1. Age group 18-65 years old
2. Both genders
3. Patients with American Society of Anesthesiologist physical status classification of 1 or 2.

Exclusion Criteria:

1. Patients who are less than 18 years old or more than 65 years old.
2. Patients with planned scheduled recovery in the intensive care unit or if more than 10 minutes had elapsed since tracheal extubation until NMB monitoring at the PACU.
3. Patients on medications that interfere with muscle activity.
4. Known allergy to neuromuscular blocking agents.
5. Pregnancy or suspected pregnancy.
6. Neuro-muscular diseases.
7. Patients refusing to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be scheduled to undergo elective surgical procedures requiring the use of neuromuscular blocking drugs.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
correlation between residual neuromuscular block risk prediction score and train of four | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No